CLINICAL TRIAL: NCT01200667
Title: uPHI: Wireless Body Area Network Core Technology
Acronym: uPHI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Ray-Jade Chen/ Deputy Superintendent, Taipei Medical University Wan Fang Hospital
Other Study IDs: 0990004864
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Asystole; Sinus Bradycardia; Sinus Tachycardia; Sinus Arrhythmia; Atril Fibrillation
MeSH Terms: conditions — Heart Arrest; Tachycardia, Sinus; Arrhythmia, Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The application scenario is shown in the figure below: the user utilizes an ECG-based wireless sensor (WiBoC Chipset), and transmit those signals to a mobile-phone device that has an embedded expert system integrated. With the aid of 3G system, a remote healthcare monitoring center receives those uploaded signals and stores into the application server. According to the events from this server, the people on service responses to the emergency and takes the corresponding process.

ELIGIBILITY:
Inclusion Criteria:

* Emergency patient with chest pain.
* Emergency patients were implementation of 12-lead EKG during observation.
* Out-patient services of Cardiology with arrhythmia history.
* Adults over 20 years old.

Exclusion Criteria:

* The patient required the intervention of resuscitation and cardiac massage.
* Chest trauma
* On pacemaker

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Emergency patient with chest pain.
  * Emergency patients were implementation of 12-lead EKG during observation.
  * Out-patient services of Cardiology with arrhythmia.
  * Adults over 20 years old.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Jade Chen, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University Wan Fang Hospital, Taipei, Taiwan